CLINICAL TRIAL: NCT01365429
Title: Novel Lung Trial: Normothermic Ex Vivo Lung Perfusion (Evlp) As An Assessment Of Extended/Marginal Donor Lungs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: XVIVO Perfusion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VSS-NA-001, XVO-NA-002
Record Dates: First submitted 2011-06-02; First posted 2011-06-03 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Lung Transplant
Keywords: Lung Transplant, Transplantation Lung
MeSH Terms: interventions — Photoelectron Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EVLP Group (Experimental): EVLP Group are those recipient lung transplant patients that received donor lungs that had been placed on the XPS™ with Steen Solution™ and undergone ex-vivo lung perfusion before being transplanted.
  Interventions: Device: XPS™ with Steen Solution™
- Control Group (No Intervention): Control Group are those recipient lung transplant patients that receive donor lungs via conventional transplant.

INTERVENTIONS:
Device: XPS™ with Steen Solution™ — The XPS™ System is an integrated cardiac bypass system comprised of various components such as a Maquet CardioHelp centrifugal pump (K102726), the HicoVariotherm Heater/Cooler, the Hamilton C2 ICU (intensive care unit) pressure- controlled ventilator (K092148), the perfusate gas monitors, and the display monitors. The XPS™ System is responsible for housing the organ for preservation, providing the normothermic environment, and perfusing the organ with the STEEN Solution™. Donor lungs that meet inclusion criteria are placed on the XPS™ and rewarmed and perfused with STEEN Solution™ and ventilated for 3-6 hours. If the lungs meet transplant suitability, they are cooled down and transplanted into a consented recipient that meet's trial criteria.
  Other Names: EVLP; ex vivo lung perfusion
  Arms: EVLP Group

SUMMARY:
Human donor lungs that do not meet the standard clinical criteria for donor lung utilization but fit into the study inclusion criteria will be retrieved from the donor using current donor lung retrieval techniques.

DETAILED DESCRIPTION:
These lungs will be brought to the study transplant center to be re-assessed by the transplant team. The lungs will be physiologically assessed during ex vivo perfusion with Steen Solution. Perfusion of these lungs will be performed using Steen solution with the addition of methylprednisolone, heparin and antibiotics. With respect to the decision of lung utilization those organs with a delta pO2 (Δ pO2 = Pulmonary vein pO2 - pulmonary artery pO2) during ex vivo perfusion assessment > 350mmHg, good lung compliance, and a favorable opinion of the transplant surgeon will be considered transplantable. Lungs will be excluded for transplantation: if the Δ pO2 is less than 350mmHg or if they demonstrate >10% deterioration in any of the following functional parameters: pulmonary vascular resistance (PVR), dynamic compliance or airway pressures. Lungs will also be excluded if they are deemed unsuitable based on the clinical judgment of the lung transplant surgeon.

ELIGIBILITY:
Recipient Inclusion/Exclusion Criteria The recipient inclusion/exclusion criteria apply to patients enrolled in the control or EVLP treatment arms.

1. Recipient Inclusion Criteria

   1. Requires single or bilateral lung transplant.
   2. Male or Female, 18 years of age or older.
   3. Subject or Subject's Representative provides a legally effective informed consent.
2. Recipient exclusion Criteria

   1. A recipient is HIV positive.
   2. A recipient has active Hepatitis.
   3. Investigator believes that the recipient has infection that excludes them from transplant in the study.
   4. To receive multi-organ transplant.
   5. Is on hemodialysis or has chronic severe renal dysfunction. Severe renal dysfunction is defined as a glomerular filtration rate of 29 or less (mL/min/1.73m2).
   6. Is to have planned concurrent cardiac procedures.
   7. A recipient is a re-transplant. (A re-transplant is defined as a recipient having the removal and transplant of a previously transplanted lung. A recipient with a previously single lung transplant is eligible to enroll in the trial if it is for the other lung and within 6 months of previous transplant.)
   8. A recipient is on Nova Lung, ECMO, or on mechanical ventilation. (CPAP and BIPAP are not exclusionary)

Donor Inclusion/Exclusion Criteria for EVLP Assessment

1. Donor Inclusion Criteria

   1. The Donor lung must meet the following criteria to proceed with EVLP:
   2. At the time of the clinical evaluation , the PaO2/FiO2 ≤ 300mmHg Or If PaO2/FiO2 > 30mmHg and the donor has any one or more of the following donor risk factors:

      * Multiple blood transfusions.
      * Pulmonary edema detected via CXR, bronchoscopy or palpation of lungs.
      * Donation after circulatory death donors.
      * Investigator evaluation of donor lung as "unsuitable" for standard criteria for lung transplant. List reason for "unsuitable" determination.
2. Donor Exclusion Criteria

   1. Lung has significant pneumonia and/or persistent purulent secretions on bronchoscopy as determined by investigator.
   2. Donor has known significant aspiration of gastric contents within the lung.
   3. Donor lung has significant mechanical lung injury or trauma determined by chest x-ray, bronchoscopy, CT Scan or visual inspection.
   4. Donor lung has active infectious disease such as HIV, Hepatitis B or C, HTLV or Syphilis. Note: This information is not available at the start of EVLP. Therefore this criteria can be assessed during or post EVLP, but prior to transplant.

Donor Inclusion/Exclusion Criteria for Transplant Suitability after EVLP

1. Donor Inclusion Criteria for Transplant Suitability

   1. Surgeon must be clinically satisfied with the lung evaluation (i.e.) overall improvement, if not, the reason for refusal must be listed.
   2. Stability or improvement of other lung function parameters during EVLP perfusion - PVR, Compliance, Airway Pressures.
   3. Two delta PO2 greater than 350 mmHg, if two delta PO2 mm Hg are not met than three out of four of the following parameters must be present:

      * One delta PO2 of > 350 or absolute PO2 of > 400.
      * Chest x-ray findings with absence or improvement of pulmonary edema/infiltrates
      * Compliance static (greater than 35 single and greater than 60 for a double)
      * Absence of consolidation by palpation
2. Donor Exclusion Criteria for Transplant Suitability after EVLP

   1. All delta PO2 (s) are less than 350 mmHg (measured with a FiO2 set at 1.0) or all absolute PO2s are less than 400.
   2. Overall greater than 10-15% Functional deterioration of other lung function across all parameters (PVR, Compliance, PawP) with chest x-ray findings showing deterioration.
   3. Donor lung positive for infectious diseases such as HIV, Hepatitis B or C, or Syphilis.

Note: This information is not available until at the start of EVLP. Therefore this criteria can be assessed during or post EVLP, but prior to transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2011-05; Primary Completion 2017-12 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
PAS Study Primary Endpoint | 3 Years
  The primary end point is a co-primary endpoint comparing survival rates and rates of grade 3 PGD at 72 hours with success if and only if both endpoints are met.
  Treatment Group (T) = EVLP transplant subjects Control Group (C) = standard transplant subjects
  Co-Primary Endpoints:
  Endpoint #1: Survival of T is non-inferior to C Ho: C - T ≥ M1 (T is inferior to the control by M1 or more) Ha: C - T < M1 (T is inferior to the control by less than M1) where M1 = 0.12 Endpoint #2: Rate of grade 3 PGD at 72 hours for T is non-inferior to the rate for C Ho: C - T ≥ M2 Ha: C - T < M2 where M2 = 0.12
PMA Study Primary Endpoint | 72hrs and Survival
  The primary end point is non-inferiority of the 3-year survival rate of the EVLP group as compared to 3-year survival rate of the control group.
  Ho: C - T ≥ M3 (T is inferior to the control by M3 or more) Ha: C - T < M3 (T is inferior to the control by less than M3) where M3 = 0.12

SECONDARY OUTCOMES:
PMA Secondary Endpoints | 3 Years
  Primary Lung Graft Dysfunction (PGD) is an indicator for significant morbidity The PMA secondary endpoints are as follows:
  * FEV1 at 3 mos, 6 mos, 9 mos, and 1 yr
  * PGD score at 24 and 48 hrs
  * ICU LOS
  * Hospital LOS
  * Use of ECMO due to lung function post transplant
  * Duration of mechanical ventilation post transplant
  * Quality of Life and functional status at one year
PAS Secondary Endpoint: | 5 Years
  Quality of Life measured by functional status, physical capability, and employment limitations.
  * Episodes of rejection per UNOS registry
  * FEV1 at 1, 2, 3, 4, and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jaya Tiwari, BS, CCRP, Study Director — XVIVO Perfusion, Inc
Locations (18):
- United States (18):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - University of Florida-Gainesville, Gainesville, Florida
  - Tampa General Hospital, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford, Detroit, Michigan
  - Barnes Jewish Hospital, St Louis, Missouri
  - Columbia University Medical Centre, New York, New York
  - Duke University, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Background] Pierre AF, Sekine Y, Hutcheon MA, Waddell TK, Keshavjee SH. Marginal donor lungs: a reassessment. J Thorac Cardiovasc Surg. 2002 Mar;123(3):421-7; discussion, 427-8. doi: 10.1067/mtc.2002.120345. PMID 11882811
- [Background] Fisher AJ, Donnelly SC, Hirani N, Haslett C, Strieter RM, Dark JH, Corris PA. Elevated levels of interleukin-8 in donor lungs is associated with early graft failure after lung transplantation. Am J Respir Crit Care Med. 2001 Jan;163(1):259-65. doi: 10.1164/ajrccm.163.1.2005093. PMID 11208654
- [Background] Power BM, Van Heerden PV. The physiological changes associated with brain death--current concepts and implications for treatment of the brain dead organ donor. Anaesth Intensive Care. 1995 Feb;23(1):26-36. doi: 10.1177/0310057X9502300107. PMID 7778744
- [Background] Avlonitis VS, Wigfield CH, Golledge HD, Kirby JA, Dark JH. Early hemodynamic injury during donor brain death determines the severity of primary graft dysfunction after lung transplantation. Am J Transplant. 2007 Jan;7(1):83-90. doi: 10.1111/j.1600-6143.2006.01593.x. PMID 17227559
- [Background] Botha P, Fisher AJ, Dark JH. Marginal lung donors: A diminishing margin of safety? Transplantation. 2006 Nov 27;82(10):1273-9. doi: 10.1097/01.tp.0000236099.52382.74. PMID 17130774
- [Background] Kawut SM, Reyentovich A, Wilt JS, Anzeck R, Lederer DJ, O'Shea MK, Sonett JR, Arcasoy SM. Outcomes of extended donor lung recipients after lung transplantation. Transplantation. 2005 Feb 15;79(3):310-6. doi: 10.1097/01.tp.0000149504.53710.ae. PMID 15699761
- [Background] Botha P, Trivedi D, Weir CJ, Searl CP, Corris PA, Dark JH, Schueler SV. Extended donor criteria in lung transplantation: impact on organ allocation. J Thorac Cardiovasc Surg. 2006 May;131(5):1154-60. doi: 10.1016/j.jtcvs.2005.12.037. PMID 16678604
- [Background] Cohen RG, Starnes VA. Living donor lung transplantation. World J Surg. 2001 Feb;25(2):244-50. doi: 10.1007/s002680020025. PMID 11338028
- [Background] Yamane M, Date H, Okazaki M, Toyooka S, Aoe M, Sano Y. Long-term improvement in pulmonary function after living donor lobar lung transplantation. J Heart Lung Transplant. 2007 Jul;26(7):687-92. doi: 10.1016/j.healun.2007.04.008. Epub 2007 Jun 13. PMID 17613398
- [Background] Steen S, Sjoberg T, Pierre L, Liao Q, Eriksson L, Algotsson L. Transplantation of lungs from a non-heart-beating donor. Lancet. 2001 Mar 17;357(9259):825-9. doi: 10.1016/S0140-6736(00)04195-7. PMID 11265950
- [Background] de Antonio DG, Marcos R, Laporta R, Mora G, Garcia-Gallo C, Gamez P, Cordoba M, Moradiellos J, Ussetti P, Carreno MC, Nunez JR, Calatayud J, Del Rio F, Varela A. Results of clinical lung transplant from uncontrolled non-heart-beating donors. J Heart Lung Transplant. 2007 May;26(5):529-34. doi: 10.1016/j.healun.2007.01.028. PMID 17449425
- [Background] Steen S, Liao Q, Wierup PN, Bolys R, Pierre L, Sjoberg T. Transplantation of lungs from non-heart-beating donors after functional assessment ex vivo. Ann Thorac Surg. 2003 Jul;76(1):244-52; discussion 252. doi: 10.1016/s0003-4975(03)00191-7. PMID 12842550
- [Background] Snell GI, Oto T, Levvey B, McEgan R, Mennan M, Higuchi T, Eriksson L, Williams TJ, Rosenfeldt F. Evaluation of techniques for lung transplantation following donation after cardiac death. Ann Thorac Surg. 2006 Jun;81(6):2014-9. doi: 10.1016/j.athoracsur.2006.01.014. PMID 16731122
- [Background] Cypel M, Sato M, Yildirim E, Karolak W, Chen F, Yeung J, Boasquevisque C, Leist V, Singer LG, Yasufuku K, Deperrot M, Waddell TK, Keshavjee S, Pierre A. Initial experience with lung donation after cardiocirculatory death in Canada. J Heart Lung Transplant. 2009 Aug;28(8):753-8. doi: 10.1016/j.healun.2009.05.009. Epub 2009 Jun 28. PMID 19632569
- [Background] Mason DP, Thuita L, Alster JM, Murthy SC, Budev MM, Mehta AC, Pettersson GB, Blackstone EH. Should lung transplantation be performed using donation after cardiac death? The United States experience. J Thorac Cardiovasc Surg. 2008 Oct;136(4):1061-6. doi: 10.1016/j.jtcvs.2008.04.023. PMID 18954650
- [Background] Orens JB, Boehler A, de Perrot M, Estenne M, Glanville AR, Keshavjee S, Kotloff R, Morton J, Studer SM, Van Raemdonck D, Waddel T, Snell GI; Pulmonary Council, International Society for Heart and Lung Transplantation. A review of lung transplant donor acceptability criteria. J Heart Lung Transplant. 2003 Nov;22(11):1183-200. doi: 10.1016/s1053-2498(03)00096-2. No abstract available. PMID 14585380
- [Background] Ware LB, Wang Y, Fang X, Warnock M, Sakuma T, Hall TS, Matthay M. Assessment of lungs rejected for transplantation and implications for donor selection. Lancet. 2002 Aug 24;360(9333):619-20. doi: 10.1016/s0140-6736(02)09774-x. PMID 12241936
- [Background] Steen S, Ingemansson R, Eriksson L, Pierre L, Algotsson L, Wierup P, Liao Q, Eyjolfsson A, Gustafsson R, Sjoberg T. First human transplantation of a nonacceptable donor lung after reconditioning ex vivo. Ann Thorac Surg. 2007 Jun;83(6):2191-4. doi: 10.1016/j.athoracsur.2007.01.033. PMID 17532422
- [Background] Ingemansson R, Eyjolfsson A, Mared L, Pierre L, Algotsson L, Ekmehag B, Gustafsson R, Johnsson P, Koul B, Lindstedt S, Luhrs C, Sjoberg T, Steen S. Clinical transplantation of initially rejected donor lungs after reconditioning ex vivo. Ann Thorac Surg. 2009 Jan;87(1):255-60. doi: 10.1016/j.athoracsur.2008.09.049. PMID 19101308
- [Background] Rega FR, Jannis NC, Verleden GM, Lerut TE, Van Raemdonck DE. Long-term preservation with interim evaluation of lungs from a non-heart-beating donor after a warm ischemic interval of 90 minutes. Ann Surg. 2003 Dec;238(6):782-92; discussion 792-3. doi: 10.1097/01.sla.0000098625.24363.d9. PMID 14631215
- [Background] Rega FR, Wuyts WA, Vanaudenaerde BM, Jannis NC, Neyrinck AP, Verleden GM, Lerut TE, Van Raemdonck DE. Nebulized N-acetyl cysteine protects the pulmonary graft inside the non-heart-beating donor. J Heart Lung Transplant. 2005 Sep;24(9):1369-77. doi: 10.1016/j.healun.2004.10.013. PMID 16143259
- [Background] Erasmus ME, Fernhout MH, Elstrodt JM, Rakhorst G. Normothermic ex vivo lung perfusion of non-heart-beating donor lungs in pigs: from pretransplant function analysis towards a 6-h machine preservation. Transpl Int. 2006 Jul;19(7):589-93. doi: 10.1111/j.1432-2277.2006.00318.x. PMID 16764638
- [Background] Egan TM, Haithcock JA, Nicotra WA, Koukoulis G, Inokawa H, Sevala M, Molina PL, Funkhouser WK, Mattice BJ. Ex vivo evaluation of human lungs for transplant suitability. Ann Thorac Surg. 2006 Apr;81(4):1205-13. doi: 10.1016/j.athoracsur.2005.09.034. PMID 16564244
- [Background] Wierup P, Haraldsson A, Nilsson F, Pierre L, Schersten H, Silverborn M, Sjoberg T, Westfeldt U, Steen S. Ex vivo evaluation of nonacceptable donor lungs. Ann Thorac Surg. 2006 Feb;81(2):460-6. doi: 10.1016/j.athoracsur.2005.08.015. PMID 16427831
- [Background] Cypel M, Yeung JC, Hirayama S, Rubacha M, Fischer S, Anraku M, Sato M, Harwood S, Pierre A, Waddell TK, de Perrot M, Liu M, Keshavjee S. Technique for prolonged normothermic ex vivo lung perfusion. J Heart Lung Transplant. 2008 Dec;27(12):1319-25. doi: 10.1016/j.healun.2008.09.003. PMID 19059112
- [Background] Cypel M, Rubacha M, Yeung J, Hirayama S, Torbicki K, Madonik M, Fischer S, Hwang D, Pierre A, Waddell TK, de Perrot M, Liu M, Keshavjee S. Normothermic ex vivo perfusion prevents lung injury compared to extended cold preservation for transplantation. Am J Transplant. 2009 Oct;9(10):2262-9. doi: 10.1111/j.1600-6143.2009.02775.x. Epub 2009 Aug 6. PMID 19663886
- [Background] Inci I, Ampollini L, Arni S, Jungraithmayr W, Inci D, Hillinger S, Leskosek B, Vogt P, Weder W. Ex vivo reconditioning of marginal donor lungs injured by acid aspiration. J Heart Lung Transplant. 2008 Nov;27(11):1229-36. doi: 10.1016/j.healun.2008.07.027. Epub 2008 Oct 1. PMID 18971096
- [Background] Yeung JC, Cypel M, Waddell TK, van Raemdonck D, Keshavjee S. Update on donor assessment, resuscitation, and acceptance criteria, including novel techniques--non-heart-beating donor lung retrieval and ex vivo donor lung perfusion. Thorac Surg Clin. 2009 May;19(2):261-74. doi: 10.1016/j.thorsurg.2009.02.006. PMID 19662970
- [Background] Van Raemdonck D, Neyrinck A, Verleden GM, Dupont L, Coosemans W, Decaluwe H, Decker G, De Leyn P, Nafteux P, Lerut T. Lung donor selection and management. Proc Am Thorac Soc. 2009 Jan 15;6(1):28-38. doi: 10.1513/pats.200808-098GO. PMID 19131528